CLINICAL TRIAL: NCT00411047
Title: A Phase II, Open Label Study of Gefitinib (IRESSA) in Treatment-Naïve Subjects With Stage IIIB or IV Non-Small Cell Lung Cancer and Somatic Activating Mutations in the Epidermal Growth Factor Receptor
Brief Title: Gefitinib in Treating Patients With Previously Untreated Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-291; IRUSIRES0483 (Other: AstraZeneca)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gefitinib — oral drug taken daily around the same time
  Other Names: IRESSA

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients with previously untreated stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective tumor response rate in patients with previously untreated stage IIIB or IV non-small cell lung cancer with somatic activating mutations in the TK region of the epidermal growth factor receptor (EGFR) gene treated with gefitinib.

Secondary

* Determine response duration, progression-free survival, and overall survival of patients treated with this drug.
* Determine the safety of this drug in these patients.
* Compare the ability of various somatic activating mutations in the TK region of the EGFR gene to predict response in patients treated with this drug.
* Compare the ability of various somatic activating mutations in the TK region of the EGFR gene to predict toxicity of this drug in these patients.
* Define a molecular profile in patients who initially respond to treatment with this drug but subsequently progress on therapy.
* Determine the significance of germline polymorphisms of the EGFR gene, somatic amplification of the EGFR gene, and other molecular factors for their association with clinical outcome parameters in these patients.

OUTLINE: This is an open-label study.

Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed non-small cell lung cancer (NSCLC)

  * No squamous cell histology
* Stage IIIB (with pleural effusion) or stage IV disease
* Must meet ≥ 1 of the following criteria:

  * Female
  * Adenocarcinoma tumor histology
  * No history of smoking, defined as smoking < 100 cigarettes (5 standard packs of cigarettes) in a lifetime, < 20 oz of pipe tobacco in a lifetime, OR < 100 cigars in a lifetime
  * Asian/Pacific Rim ethnicity, defined as Japanese, Chinese, Korean, or other Asian/Pacific Rim ethnicity
* Must have activating mutations in the TK region of the epidermal growth factor receptor (EGFR) gene
* Measurable disease
* No symptomatic or newly diagnosed CNS metastases that have not been definitively treated with radiotherapy and/or surgery

  * History of CNS metastases or cord compression allowed if definitively treated and clinically stable

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (5 times ULN if liver has tumor involvement)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known severe hypersensitivity to gefitinib or any other component of gefitinib tablets
* No evidence of clinically active interstitial lung disease

  * Patients with chronic, stable radiographic changes who are asymptomatic are eligible
* No other concurrent malignancy or malignancy diagnosed within the past 5 years except for basal cell carcinoma of the skin or cervical cancer in situ
* No concurrent severe or uncontrolled systemic disorder
* No evidence of any other significant clinical disorder or laboratory finding that, in the opinion of the investigator, would preclude study participation
* Able to tolerate protocol treatment, in the opinion of the investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy, biological therapy, immunotherapy, or hormonal therapy for NSCLC, including adjuvant and neoadjuvant treatment
* No prior radiotherapy to the target lesion

  * Prior radiotherapy to bony disease or CNS disease allowed
* At least 2 weeks since prior radiotherapy and recovered
* More than 30 days since prior non-FDA approved or investigational agents
* No prior EGFR antagonists
* At least 2 weeks since prior and no concurrent phenytoin, carbamazepine, rifampin, barbiturates, or Hypericum perforatum (St. John's wort)
* No concurrent chemotherapy, immunotherapy, hormonal therapy, nonpalliative radiotherapy, surgery for cancer, or other experimental medications
* No other concurrent specific antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate

SECONDARY OUTCOMES:
Response duration, progression-free survival, and overall survival
Safety
Ability of various somatic activating mutations in the TK region of the epidermal growth factor receptor (EGFR) gene to predict response and toxicity
Molecular profile
Significance of germline polymorphisms of the EGFR gene, somatic amplification of the EGFR gene, and other molecular factors for their association with clinical outcome parameters

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials